CLINICAL TRIAL: NCT00960180
Title: A Study Investigating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ascending Single Doses of Orally Administered MR1817 in Healthy Adult Subjects
Brief Title: Study Evaluating Single Ascending Doses of MR1817
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 3260A1-1000
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2011-05

CONDITIONS: Adult

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MR1817
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MR1817
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This is a first-in-human study of MR1817. This study will provide an initial assessment of the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of MR1817 after administration of ascending single oral doses to healthy adult subjects.

ELIGIBILITY:
Inclusion criteria: 1- Men or women of non-childbearing potential (WONCBP) aged 18 to 55 years inclusive at screening.

2- Body mass index (BMI) in the range of 18 to 32 kg/m2 and body weight ≥50 kg. 3- Healthy as determined by the investigator on the basis of screening evaluations.

Exclusion criteria: 1- Presence or history of any disorder that may prevent the successful completion of the study. 2- Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease. 3- History of drug abuse within 1 year before study day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety based on adverse event reporting, physical examinations, vital sign evaluations, 12-lead ECGs and routine laboratory tests | 6 weeks

SECONDARY OUTCOMES:
MR1817 plasma and urine concentration. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miller, Study Director — Fulcrum Pharma (Europe) Ltd
Locations (1):
- Cambridge, United Kingdom